CLINICAL TRIAL: NCT05465785
Title: A Clinical Trial to Evaluate the Immunogenicity Bridging Between Different Manufacture Scales of Recombinant COVID-19 Vaccine (Sf9 Cell) in Healthy Population Aged 18-59 Years
Brief Title: A Clinical Trial of Immuno-bridging Between Different Manufacture Scales of Recombinant COVID-19 Vaccine (Sf9 Cell)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT141
Record Dates: First submitted 2022-02-13; First posted 2022-07-20 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2 Pneumonia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot batch (Experimental): Three doses of Recombinant COVID-19 vaccine (Sf9 cell) at the schedule of day 0, 21，42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cell)
- Commercial batch (Active Comparator): Three doses of Recombinant COVID-19 vaccine (Sf9 cell) at the schedule of day 0, 21，42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cell)

INTERVENTIONS:
Biological: Recombinant COVID-19 vaccine (Sf9 cell) — This vaccine is made by using baculovirus as a vector and expressing SARS-CoV-2 S-RBD in Sf9 cells, which is purified

SUMMARY:
This is a randomized, double-blind , non-inferiority design study, to evaluate the Immunogenicity bridging between different manufacture scales of Recombinant COVID-19 Vaccine (Sf9 Cell) in healthy population aged 18-59 years with immunization procedures 0, 21, 42 days .

DETAILED DESCRIPTION:
This is a randomized, double-blind , non-inferiority design study, to evaluate the Immunogenicity bridging between different manufacture scales of Recombinant COVID-19 Vaccine (Sf9 Cell) in healthy population aged 18-59 years with vaccination course 0, 21, 42 days. 892 subjects aged 18-59 years are recruited and randomly inoculated in a 1:1 ratio from a pilot or commercial batch of Recombinant COVID-19 Vaccine (Sf9 Cell).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 18-59 years.
* Signed informed consent forms of the subjects have been obtained.
* Able and willing to comply with the requirements of the clinical trial protocol and able to complete approximately 8 months of study follow-up.
* Axillary temperature < 37.3℃. Subjects who fulfill all the required conditions for receiving the candidate vaccine as established by medical history and physical examination and determined by investigators.

Exclusion Criteria:

* Positive SARS-CoV-2 antibodies (IgG or IgM) screening results.
* Positive SARS-CoV-2 Antigen screening results.
* History of COVID-19 vaccination.
* Previously diagnosed with COVID-19 infection.
* History of HIV infection.
* History or family history of convulsion, epilepsy, encephalopathy and psychosis.
* Allergy to any component of the candidate vaccine, severe allergy to vaccine in the past, and history of allergy.
* Women with positive urine pregnancy test results, pregnant, lactating women, or women who have a pregnancy plan during the study.
* Patients with acute febrile diseases and infectious diseases.
* Patients with a history of SARS.
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension that cannot be controlled by drugs, etc.
* Serious chronic diseases or progressive stage of a disease that cannot be steadily controlled, such as asthma, diabetes mellitus, thyroid disease, etc.
* Congenital or acquired angioedema/angioneurotic edema.
* Urticaria 1 year before receiving the candidate vaccine.
* Asplenia or functional asplenia.
* Thrombocytopenia or other coagulation disorders (which may contraindicate intramuscular injection).
* Fear of needles.
* Any immunosuppressant, antiallergic therapy, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) in the past 6 months.
* Blood products within 4 months prior to receiving the candidate vaccine.
* Any other investigational medicine(s) within 1 month prior to the candidate vaccine.
* Any live attenuated vaccine within 1 month prior to the candidate vaccine.
* Any subunit vaccine or inactivated vaccine within 14 days prior to the candidate vaccine.
* Receiving antituberculosis treatment.
* Medical, psychological, social or other factors, which in the discretion of the investigators fail to meet the requirements in the trial protocol or affect the subjects to sign the ICFs.

Exclusion criteria for the second/third dose:

In this trial, the second/third vaccination may be stopped in some cases. They include systemic allergic reaction, severe hypersensitivity, or intolerable Grade 3 or above ARs after the previous dose of vaccine. If these reactions occur, the subjects should not continue to receive the second/third vaccination.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse reactions(ARs). | Day 0 to day 7
  The incidence of ARs within 7 days after each vaccination.
Anti-SARS-CoV-2 specific neutralizing antibodies expressed as geometric mean titer (GMT)and seroconversion rate (SCR). | Day 72
  The GMT and SCR of anti-SARS-CoV-2 specific neutralizing antibodies (euvirus) of the subjects on day 30 after the third vaccination.

SECONDARY OUTCOMES:
The incidence of ARs. | Day 0 to Day 72
  The incidence of ARs from Day 0 to Day 72.
The incidence of adverse events (AEs). | Day 0 to Day 72
  The incidence of adverse events (AEs) from Day 0 to Day 72.
The incidence of serious adverse events (SAEs). | Day 0 to 6 months after the third vaccination.
  The incidence of SAEs from day 0 through 6 months after the third vaccination.
The Geometric Mean Fold Increase (GMI) of the anti-SARS-COV-2 specific neutralizing antibody. | Day 72
  The GMI of the anti-SARS-COV-2 specific neutralizing antibody of the subjects on day 30 after the third vaccination.
The Geometric Mean Titre (GMT), Seroconversion Rate (SCR) and GMI of anti-SARS-COV-2 S-RBD Immunoglobulin (IgG) antibody | Day 72
  The GMT, SCR and GMI of anti-SARS-COV-2 S-RBD IgG antibody of the subjects on day 30 after the third vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Huai'an, Jiangsu, China